CLINICAL TRIAL: NCT06159283
Title: Intravenous Immunoglobulin Replacement Therapy for Persistent COVID-19 in Patients With B-cell Impairment: a Multicenter Randomized Controlled Trial
Brief Title: Intravenous Immunoglobulin Replacement Therapy for Persistent COVID-19 in Patients With B-cell Impairment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jaehoon Ko (Other)
Responsible Party: Sponsor-Investigator, Jaehoon Ko, Assistant Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-11-078
Record Dates: First submitted 2023-12-04; First posted 2023-12-06 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Immunoglobulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVIG administration (Experimental): The patients who will meet the inclusion criteria will be administered IVIG at a dose of 1,000 mg/kg, divided over 2-3 days. After administration, the patient's condition will be thoroughly observed. In case of adverse effects from an increased administration rate, the rate will be reduced immediately or suspended until symptom improvement. Other standards of care can be continued.
  Interventions: Drug: Immunoglobulins
- Standard Of Care (No Intervention): The same anti-viral, anti-inflammatory, and anti-coagulation treatment criteria are applied to the treatment group. If the primary endpoint will be not reached by day 14 of randomization, IVIG can be given at a dose of 1,000 mg/kg based on clinicians' discretion.

INTERVENTIONS:
Drug: Immunoglobulins — Dosage is Immunoglobulin 1,000mg/kg IV. It administer over 2~3 days.
  Other Names: Immunoglobulins in this study uses commercially avilable drug.
  Arms: IVIG administration

SUMMARY:
This is a multicenter, randomized controlled trial aiming to investigate the efficacy of intravenous immunoglobulin (IVIG) replacement therapy under the hypothesis that immunoglobulin replacement would have therapeutic effects on persistent COVID-19 in patients with B-cell impairment.

DETAILED DESCRIPTION:
This project aims to provide passive immunization to patients with persistent COVID-19 who experience inflammation owing to continuous replication of SARS-CoV-2, as a consequence of B-cell impairment that hinders normal antibody formation. As opposed to relying on the non-specific immune mechanism of IVIG in other studies, this trial focuses on the antiviral effect and antibody-dependent cytotoxicity induced by SARS-CoV-2-specific antibodies from plasma donors who have formed high antibody titers through vaccination and breakthrough infections. Thus, in contrast to previous studies, the therapy may demonstrate clinical efficacy. In this work, we aim to elucidate the role of IVIG in treating persistent COVID-19 in patients with B-cell depletion who cannot produce antibodies, and to establish grounds for clinical application of the therapy.

Once the participants voluntarily provide written consent to participate in the trial, they will undergo screening tests, and eligible participants will be randomly assigned to the treatment or control (standard of care) group in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written consent to participate in the trial
2. Age≥ 19 years
3. Diagnosed as COVID-19: the definitive diagnosis of COVID-19 will be made at a healthcare facility based on COVID-19 tests approved in Korea, such as reverse transcription polymerase chain reaction (RT-PCR), Xpert, film array, and rapid antigen test (RAT).
4. The diagnosis of persistent COVID-19 will be made following the criteria below:

<!-- -->

1. No improvement or worsening of symptoms/signs of active inflammation, such as fever, pneumonia, and dyspnea requiring oxygen, even after 2 weeks of the initial symptom onset or diagnosis of COVID-19 (persisting symptoms/signs at or after the third week of illness).
2. The day count for the disease course is based on the symptom onset or diagnosis date, whichever is earlier, with Day 1 being the date of symptom onset or diagnosis. The third week refers to the period including and following Day 15. For the purpose of day count calculation, self-test results using RAT are accepted.
3. Both symptoms and signs indicative of active inflammation must be present. This status corresponds to the Modified WHO clinical progression scale of ≥ 4.

   * Symptoms include at least one of the following.

     1. Fever of 37.8°C or higher lasting for >48 h (determined based on self-measurement and statements from the patient or caregiver, with fevers persisting from Day 13 to Day 15 also accepted)
     2. Persistent cough despite taking appropriate expectorants and cough suppressants
     3. Dyspnea upon walking on a flat surface (modified Medical Research Council grade >2) ② At least one of the following signs of active inflammation must be present.

     <!-- -->

     1. Pulmonary infiltration suggestive of COVID-19 observed in chest radiograph or computed tomography scan findings. Findings may vary, from ground-glass opacities to patchy consolidation, and are determined by the clinician or radiologist.
     2. Decreased oxygen saturation (PaO2/FiO2 ≤300 mmHg, SpO2 ≤92%, or PaO2 ≤63%) 5. Cases of patients with B-cell impairment:

(1) Patients with B-cell lineage hematologic malignancies, such as B-cell lymphoma or multiple myeloma, who are presumed to have impaired B-cell function owing to B-cell targeting chemotherapy (i.e., those receiving rituximab, CAR-T, Bispecific T-cell engager therapies), or second-line or higher treatments, such as autologous stem cell transplantation (AutoPBSCT) (2) Patients suffering from diseases known to result in B-cell depletion, such as Good's syndrome associated with thymoma (3) Cases of patients with a congenital primary immunodeficiency who have reduced antibody formation and have not undergone IVIG replacement in the past 3 months.

Among these, those who received B-cell targeting chemotherapy within the past 3 months are eligible for enrollment based on clinical criteria, but other patients must confirm the reduction of peripheral B cells to <1% via flow cytometry to be eligible for enrollment.

Exclusion Criteria:

1. Difficulty controlling the underlying disease or life expectancy of <3 months even after COVID-19 is successfully treated.
2. T-cell impairment.

(1)T-cell suppressive drugs (e.g., cyclosporine, tacrolimus) cannot be suspended owing to organ transplantation or autoimmune disorder.

(2) Patients with human immunodeficiency virus (HIV) infection with a CD4 T-cell count <500 cells/μL or persistent detection of HIV viral RNA in the blood.

3. IVIG or COVID-19 convalescent plasma therapy within 3 months of screening 4. History of serious reaction or hypersensitivity to blood, blood products, blood-derived products, IVIG, and IgG 5. Immunoglobulin A (IgA) deficiency or IgA antibodies present 6. Uncontrolled hypertension (systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg) 7. Hemolytic anemia, hemorrhagic anemia 8. Impaired cardiac function [New York Heart Association Functional Class Ⅲ or IV] 9. High risk for thrombosis/embolism clinically owing to a history of cerebrovascular and cardiovascular disorders, thrombosis, or embolism 10. Cases of pregnant or breastfeeding women 11. Current participation in another clinical trial related to COVID-19 drugs 12. Cases of participants that are inappropriate to participate in the trial based on the investigator's discretion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of clinical effectiveness | 14day
  Clinical recovery

SECONDARY OUTCOMES:
Evaluation of clinical effectiveness | 30day and 60day
  Clinical recovery

CONTACTS AND LOCATIONS:
Overall Officials: Jaehoon Ko, Ph,MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Jaehoon Ko, Seoul, South Korea